CLINICAL TRIAL: NCT03600064
Title: Misoprostol for Cervical Ripening Before Copper Intrauterine Device Removal in Women Delivered Only by Elective Cesarean Section
Brief Title: Misoprostol for Cervical Ripening Before Copper Intrauterine Device Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIUD
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Intrauterine Device
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol group (Other)
  Interventions: Drug: Misoprostol
- NO intervention (No Intervention)

INTERVENTIONS:
Drug: Misoprostol — the women will be received two tablets of misoprostol 400 mcg vaginally before IUD removal (Misotac®; Sigma Pharma, SAE, Egypt).
  Arms: Misoprostol group

SUMMARY:
Intrauterine devices are the most common used method of contraception in the world, mostly in developing countries, because they offer long-term, reversible and relatively safe contraception. At present, 50% of intrauterine devices users are women of reproductive age and most of them are requesting Intrauterine device removal to regain their fertility. In general, an intrauterine device should be removed during menses or preferably immediate after menses because intrauterine device removal is usually easy because the cervix is still soft.

The intrauterine device is usually removed by firmly grasping the threads at the external os; traction should be applied away from the cervix. If resistance is present, the removal should be stopped until it is determined why the intrauterine device is not moving. Some deeply embedded intrauterine device may need to be removed by hysteroscope [4].

In practice, many women, however, have an intolerable pain during intrauterine device removal and some of them requesting painkiller or even anesthesia to allow the physician to remove it. Cervical hardening and adhesions are the major factors making IUD removal difficult especially in post-menopausal women.

Insertion and removal of IUD in nulliparous women is possible but it may carry more pain, more difficulty than in parous women. We think that this problem is also present in women has no vagina delivery before. So, the intrauterine device removal actually has some difficulty or pain in the nulliparous women, women delivered by elective caesarian section or postmenopausal women.

Many medical agents for cervical ripening prior to the removal have been emerged like misoprostol. Misoprostol is commonly used for cervical ripening in the first and second trimester miscarriage and prior intrauterine devices insertion. The use of vaginal misoprostol before intrauterine device insertion in women who had never delivered vaginally before may increase the ease and success of insertion with pain felt during the procedure .

However and up to our knowledge; no studies had been reported the effect of misoprostol on removal pain in women delivered only by elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years
2. Menstruating women
3. Nonpregnant women
4. Delivered before only by elective cesarean section
5. Women who did not receive any analgesics in the 24 h prior to Intrauterine device removal.
6. Using copper 380 A Intrauterine device for contraception only
7. Requesting Intrauterine device removal for returning of fertility

Exclusion Criteria:

1. Women with allergy to misoprostol or any medical disease that contraindicates its use
2. Ultrasonographic evidence of displaced Intrauterine device.
3. Women who will refuse to participate in the study.
4. Women who had any other type of Intrauterine device.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain perception immediate after intrauterine device removal measured by Visual analogue scale | 1 minute
  visual analogue scale from 0 to 10 score (0 means no pain, 10 means maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided